CLINICAL TRIAL: NCT00037154
Title: Saw Palmetto Extract In Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5 R01 DK056199 (completed); 5R01DK056199 (NIH)
Record Dates: First submitted 2002-05-16; First posted 2002-05-17 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia; Herbal Therapies; Complementary and Alternative Medicine; Men's Health
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — saw palmetto extract

INTERVENTIONS:
Drug: Saw Palmetto

SUMMARY:
The purpose of this study is to test whether an extract of the saw palmetto plant is effective for relieving symptoms of Benign Prostatic Hyperplasia (BPH).

DETAILED DESCRIPTION:
This proposal describes a double-blind, placebo-controlled randomized clinical trial of the effect of saw palmetto extract on symptoms, objective parameters of disease severity, and quality of life in men with moderate-to-severe benign prostatic hyperplasia. BPH, one of the most common morbid medical conditions in middle-aged and elderly men, is generally treated with alpha-adrenergic blocking agents, finasteride, surgical interventions, or no specific therapy ("watchful waiting"). In the past several years, however, many patients have begun to self-medicate with an extract of the saw palmetto plant (Serenoa repens), a medicinal herb grown in the southeastern United States. Saw palmetto has become the fifth leading medicinal herb consumed in the U.S. and is considered first-line therapy for BPH in several Western European countries. Several small studies suggest that saw palmetto may have clinical benefit, but the methodologic quality of most prior studies has been poor. Very few side effects of the herb have been observed, but few studies have been conducted for more than three months. We propose to conduct a high-quality clinical trial of saw palmetto, with careful attention to the methodologic deficiencies of prior studies. After a single-blind placebo run-in period, 224 patients with mode moderate-to-severe BPH (American Urological Association Symptom Index score greater than or equal to 8) and objective measurement of urinary obstruction, will be randomized to receive either 160mg BID of the herbal extract or an identical placebo. Patients will discontinue any other medical therapy for BPH prior to enrollment and all participants will undergo a trans-rectal ultrasound examination at baseline and closeout. Participants in the trial will be seen at 3-month intervals for a total one-year follow-up. Outcome measurements include changes in the AUASI score (the primary outcome measurement), the peak urinary flow rate, the post-void residual urine volume, the BPH Impact Index, the Olmstead County Study Questionnaire of BPH-specific symptoms and quality of life, and the Short-Form 36 (a generic health status instrument). Numerous laboratory parameters will measured at intervals throughout the trial and symptomatic side effects will be assessed.

ELIGIBILITY:
Eligibility Criteria:

* Participants must be men, aged 50 years or older with moderate-to-severe BPH.
* Participants must not have a history of prostate cancer, prior surgery on the prostate, kidney failure, or taking furosemide (Lasix), warfarin (Coumadin), or hormone medications. Individuals taking medicine for their BPH must stop them for one month (prazosin, terazosin (Hytrin), doxazosin (Cardura), tamsulosin (Flomax)) or six months (saw palmetto, finasteride (Proscar or Rogaine)) prior to entering the study.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224
Dates: Start 1999-08; Study Completion 2002-12

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Avins, MD, MPH, Principal Investigator — Northern California Kaiser Permanente; University of California, San Francisco; San Francisco Veterans Affairs Medical Center; Stephen Bent, MD, Study Director — University of California, San Francisco; San Francisco Veterans Affairs Medical Center
Locations (2):
- United States (2):
  - Northern California Kaiser Permanente, Oakland, California
  - Veterans Affairs Medical Center, San Francisco, California

REFERENCES:
- [Result] Bent S, Kane C, Shinohara K, Neuhaus J, Hudes ES, Goldberg H, Avins AL. Saw palmetto for benign prostatic hyperplasia. N Engl J Med. 2006 Feb 9;354(6):557-66. doi: 10.1056/NEJMoa053085. PMID 16467543
- [Derived] Avins AL, Bent S, Padula A, Staccone S, Badua E, Goldberg H. Initial experience with a group presentation of study results to research participants. Trials. 2008 Mar 21;9:16. doi: 10.1186/1745-6215-9-16. PMID 18355417